CLINICAL TRIAL: NCT07345585
Title: Probiotics for Autism Spectrum Disorders: a Randomized Controlled Trial (The PASD Study)
Acronym: PASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, MD,PhD,Prof, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 38/2023
Record Dates: First submitted 2025-12-09; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Lactobacillus rhamnosus GG
  Interventions: Other: Lactobacillus rhamnosus GG
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Lactobacillus rhamnosus GG — Lactobacillus rhamnosus GG
  Arms: Probiotic
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Autism spectrum disorders (ASD) are a group of severe neurodevelopmental conditions characterized by impaired communication and social interaction, as well as repetitive/stereotyped behaviors deriving from a combination of genetic and environmental factors. The ASD diagnosis rates increased dramatically over the past number of decades. The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) describes a worldwide prevalence of approximately 1%. The prevalence of ASD is 1 in 59 individuals in the US reported by the Centers for Disease Control and Prevention. According to the latest data from the Italian National Observatory for ASD, the actual prevalence in Italy is about 1/77 for children aged between 7 and 9 years, with a 4.4 times higher prevalence in male. The origin of ASD is still largely undefined. It has been hypothesized a possible role for the influence of early life alteration of gut microbiome (GM). We demonstrated an imbalance in Bacteroidetes and Firmicutes phyla with a decrease in Bacteroidetes/Firmicutes ratio in the GM of pediatric patients affected by ASD. Similar data have been observed by others. Data from ASD animal model confirm the presence of GM dysbiosis with significant correlation with behavioral, gastrointestinal and immunologic alterations. Altogether these data support the hypothesis that GM dysbiosis could be involved in the ASD pathogenesis. The ASD children present an increased prevalence of functional gastrointestinal disorders (FGIDs), mainly chronic constipation, functional diarrhea, and irritable bowel syndrome (IBS). A role for GM has been suggested also for these conditions. The presence of these disorders negatively influence the disease severity and the parental quality of life of ASD children. Starting from all these considerations GM is becoming a possible target of intervention for pediatric ASD. Probiotics are one of the most investigated strategy for a beneficial modulation of GM. Probiotics are commonly defined as live microorganisms which when ingested in adequate amounts confer a beneficial effect on the host. The most used probiotics in the pediatric age are Saccharomyces and Lactobacillus strains including Lactobacillus rhamnosus GG (LGG). Data report a beneficial influence elicited by LGG on GM structure and function. This probiotic resulted also effective in treating FGIDs patients. Preliminary evidence suggest the potential efficacy of probiotics for FGIDs treatment in ASD children. Altogether these evidence strongly support the hypothesis that LGG could exert a beneficial action in ASD children. The purpose of this study is to evaluate the therapeutic efficacy of LGG on FGIDs in ASD children.

ELIGIBILITY:
Inclusion Criteria:

* children aged 4-12 years
* children of both sex
* children with a sure diagnosis of ASD and presence of FGIDs with a GSI ≥7 from at least 3 months.

Exclusion Criteria:

* children aged <4 or >12 years
* uncertain ASD and/or FGIDs diagnosis
* FGIDs duration lasting <3 months
* concomitant presence of other chronic conditions (adverse food reactions; genetic and metabolic disorders; malformations of GI, respiratory or urinary tract; neurologic diseases; immunodeficiencies; diabetes; cardiovascular diseases; autoimmune diseases; chronic infections; chronic respiratory, GI or urinary tract diseases; obesity; tumors; malnutrition).
* use of antibiotics and/or pre-/pro-/ synbiotics during the 6 months prior to enrolment
* participation into other clinical trials during the last 12 months.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional gastrointestinal disorders (FGIDs) severity | At 16 weeks of treatment
  Severity index of gastrointestinal symptoms (GI Severity Index, GSI) - Minimum Score: 0 (Indicates absence of gastrointestinal symptoms or optimal bowel regularity) Maximum Score: 17 (Represents the highest severity of symptoms reported in the questionnaire)

SECONDARY OUTCOMES:
Kinetics of Lactobacillus rhamnosus GG (LGG) | At baseline and at 4 weeks, 8 weeks and 12 weeks of treatment
  Using the GI Severity Index (GSI) - Minimum Score: 0 (Indicates absence of gastrointestinal symptoms or optimal bowel regularity) Maximum Score: 17 (Represents the highest severity of symptoms reported in the questionnaire)
Duration of the LGG impact on FGIDs | At baseline and at 4 weeks and 12 weeks from the end of treatment
  Changes in the GSI - Minimum Score: 0 (Indicates absence of gastrointestinal symptoms or optimal bowel regularity) Maximum Score: 17 (Represents the highest severity of symptoms reported in the questionnaire)
Gut Microbiome (GM) composition | At baseline and at 16 weeks of treatment
  Shotgun metagenomics analysis
GM function: fecal short chain fatty acids (SCFAs) levels | At baseline and at 16 weeks of treatment
  Gas chromatograph(GC)-mass spectrometry (MS) analysis
ASD children behavior | At baseline, at 4 weeks, at 8 weeks, at 12 weeks and at 16 weeks of treatment, and at 4 weeks and 12 weeks from the end of treatment
  Aberrant Behavior Checklist (ABC) questionnaire - Minimum Score: 0 (Indicates the complete absence of aberrant or problematic behaviors in the assessed areas, e.g., aggression, social withdrawal, stereotypies, etc.) Maximum Score: 174 (Represents the highest severity and frequency of problematic behaviors reported in the test. All listed aberrant behaviors-such as self-injury, severe hyperactivity, complete social withdrawal, and repetitive speech-are present at maximum intensity.)
Parental quality of life | At baseline, at 4 weeks, at 8 weeks, at 12 weeks and at 16 weeks of treatment, and at 4 weeks and 12 weeks from the end of treatment
  EUROHIS QOL-8 questionnaire - Minimum Score: 8 (Indicates the lowest level of satisfaction and quality of life) Maximum Score: 40 (Indicates the highest level of satisfaction and quality of life)
Body weight | At baseline, at 4 weeks, at 8 weeks, at 12 weeks and at 16 weeks of treatment, and at 4 weeks and 12 weeks from the end of treatment
  Body weight will be evaluated in kilograms
Height | At baseline, at 4 weeks, at 8 weeks, at 12 weeks and at 16 weeks of treatment, and at 4 weeks and 12 weeks from the end of treatment
  Body weight will be evaluated in cm
Infectious diseases | At 4 weeks, at 8 weeks, at 12 weeks and at 16 weeks of treatment, and at 4 weeks and 12 weeks from the end of treatment
  It will be assessed the number of infectious episodes, type of infectious diseases, need for drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No